CLINICAL TRIAL: NCT04220151
Title: Epigenetic Changes in Hepatocellular Carcinoma Developed After Direct Acting Antiviral Therapy for Chronic Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Hepatocellular carcinoma
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Epigenetics; DNA methylation; Direct-acting antivirals
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hepatocellular carcinoma: Sixty patients with HCC
  Interventions: Genetic: DNA methylation
- Hepatic cirrhosis: Thirty patients with hepatic cirrhosis
  Interventions: Genetic: DNA methylation
- Healthy controls: Ten healthy controls.
  Interventions: Genetic: DNA methylation

INTERVENTIONS:
Genetic: DNA methylation — DNA methylation will be measured by real time polymerase chain reaction

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common type of liver cancer, its survival rate ranks only second to lung cancer and it is a severe threat to human health.

In Egypt, HCC constitutes a significant public health problem. Where it is responsible for 33.63% and 13.54% of all cancers in males and females respectively. It has a poor prognosis after discovery, which is usually at a late stage of disease. This had been strongly linked to the hepatitis C virus epidemic that affected around 10-15% of the Egyptian population during the last 3 decades, and was reported as the highest prevalence of HCV in the world. However, the pathophysiological mechanisms involved remain unclear. The occurrence of HCC is a complicated process involving multiple genes and steps. Imbalances in cellular signal transduction pathways, deficiencies in DNA repair regulating genes, activation of protooncogenes, inactivation of tumor suppressor genes and epigenetic modifications all promote the occurrence of liver cancer.

DETAILED DESCRIPTION:
HCC is the fourth leading cause of cancer mortality in 2018. The alarming incidence of HCC is explained by genetic and epigenetic alterations, as well as by the presence of risk factors: hepatitis C virus (HCV), hepatitis B virus (HBV) infection, alcohol consumption, smoking, diabetes, dietary exposure to aflatoxins, and obesity.

The development of direct-acting antivirals (DAAs) with cure rates of higher than 90% has been a major breakthrough in the management of patients with chronic HCV infection. However, although viral cure decreases the overall HCC risk in HCV-infected patients, it does not eliminate virus-induced HCC risk, especially in patients with advanced fibrosis. Furthermore, convenient biomarkers to robustly predict HCC risk after viral cure and strategies for HCC prevention are absent. These unexpected findings pose new challenges for patient management. Meanwhile, recent studies in patients treated with interferone-free therapy have also identified several risk factors for developing HCC after achieving sustained virological response (SVR), namely advanced hepatic fibrosis and higher levels of alpha feto protein and agglutinin-positive Mac-2 binding protein.

Epigenetics refers to inherited altered gene expression without an alteration of the DNA sequence itself. Epigenetic alterations, such as DNA hypomethylation or hypermethylation and aberrant expression of micro-RNAs have been studied and associated with HCC. Epigenetic changes may represent diagnostic and prognostic biomarkers of HCC.

ELIGIBILITY:
Inclusion Criteria:

* HCC treated with DAAs drugs for chronic hepatitis C in Assiut University Hospital.

Exclusion Criteria:

* Cases who started treatment for HCC like alcohol ablation or chemoembolization
* Hepatitis B infection
* Non-responder patients to DAAs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentages of methylation of DNA in patients with HCC | Baseline
  Hypermethylation is known to be associated with decreased gene expression

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar-Medina M, Avendano-Felix M, Lizarraga-Verdugo E, Bermudez M, Romero-Quintana JG, Ramos-Payan R, Ruiz-Garcia E, Lopez-Camarillo C. SOX9 Stem-Cell Factor: Clinical and Functional Relevance in Cancer. J Oncol. 2019 Apr 1;2019:6754040. doi: 10.1155/2019/6754040. eCollection 2019. PMID 31057614
- [Background] Cozma A, Fodor A, Vulturar R, Sitar-Taut AV, Orasan OH, Muresan F, Login C, Suharoschi R. DNA Methylation and Micro-RNAs: The Most Recent and Relevant Biomarkers in the Early Diagnosis of Hepatocellular Carcinoma. Medicina (Kaunas). 2019 Sep 19;55(9):607. doi: 10.3390/medicina55090607. PMID 31546948
- [Background] Saleh DA, Amr S, Jillson IA, Wang JH, Crowell N, Loffredo CA. Preventing hepatocellular carcinoma in Egypt: results of a Pilot Health Education Intervention Study. BMC Res Notes. 2015 Aug 29;8:384. doi: 10.1186/s13104-015-1351-1. PMID 26319021
- [Background] Perez S, Kaspi A, Domovitz T, Davidovich A, Lavi-Itzkovitz A, Meirson T, Alison Holmes J, Dai CY, Huang CF, Chung RT, Nimer A, El-Osta A, Yaari G, Stemmer SM, Yu ML, Haviv I, Gal-Tanamy M. Hepatitis C virus leaves an epigenetic signature post cure of infection by direct-acting antivirals. PLoS Genet. 2019 Jun 19;15(6):e1008181. doi: 10.1371/journal.pgen.1008181. eCollection 2019 Jun. PMID 31216276